CLINICAL TRIAL: NCT01350986
Title: Efficacy of Cognitive-Behavioral Based Guided Self-Help for Parents of Children With Externalizing Problem Behavior
Brief Title: Guided Self-Help for Parents of Children With Externalizing Problem Behavior
Acronym: FLOH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Research Foundation (Other)
Responsible Party: Manfred Döpfner, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DO 620/5-1; Köln Fortune (Other Grant/Funding Number: 28/2010)
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Oppositional Defiant Disorder; Attention Deficit Hyperactivity Disorders; Attention Deficit and Disruptive Behavior Disorders
Keywords: Controlled Clinical Trials, Randomized
MeSH Terms: conditions — Oppositional Defiant Disorder; Attention Deficit Disorder with Hyperactivity; Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Directive (Experimental)
  Interventions: Behavioral: Cognitive-Behavioral Self-help Workbook + Counseling Telephone Calls
- Non-Directive (Active Comparator)
  Interventions: Behavioral: Non-Directive Self-Help Workbook + Counseling Telephone Calls

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Self-help Workbook + Counseling Telephone Calls — In intervention period of 5 months parents work through 8 cognitive-behavioral self-help booklets (FLOH) and additionally receive 10 counseling telephone calls. Primary purpose of telephone calls is to clarify content of the booklets and support parents in managing their homework assignments accompanied with each booklet. 3 and 6 months after intervention period has ended, two additional booster telephone calls are provided. The booklets are based on the therapy manual "Treatment program for children with hyperactive and oppositional problem behavior (THOP)" (Döpfner, Schürmann, & Frölich, 2007) and the parent self-help book "Wackelpeter and Trotzkopf: Help for parents of children with hyperkinetic and oppositional behavior" (Döpfner, Schürmann, & Lehmkuhl, 2006).
  Other Names: FLOH
  Arms: Directive
Behavioral: Non-Directive Self-Help Workbook + Counseling Telephone Calls — In intervention period of 5 months parents are provided 8 non-directive self-help booklets and additionally receive 10 non-directive counseling telephone calls. If the telephone calls are used to clarify content of the booklets or to discuss other child and parenting related topics is at the parents' discretion. Main focus for counselor is to be congruent, empathic and to have unconditional positive regard toward the parents. 3 and 6 months after intervention period has ended, two additional booster telephone calls are provided. The booklets are based on "Parent effectiveness training" (Gordon, 1970) and "Teaching children self-discipline at home and at school" (Gordon, 1989).
  Other Names: "Parent effectiveness training"; "Teaching children self-discipline at home and at school"
  Arms: Non-Directive

SUMMARY:
The efficacy of cognitive-behavioral based guided self-help for parents of children with externalizing problem behavior is tested in a randomized clinical trial. Parents work through cognitive-behavioral self-help booklets and additionally receive counseling telephone calls every two weeks. In the control condition parents are provided non-directive self-help booklets and additionally receive counseling telephone calls. It is hypothesized that the cognitive-behavioral treatment is superior.

ELIGIBILITY:
Inclusion Criteria:

* Child diagnosis of ODD and/or ADHD based on DCL-ODD and DCL-ADHD respectively

Exclusion Criteria:

* Child IQ is below 80
* Child has diagnosis of pervasive developmental disorder (PDD)
* Indication for inpatient/intensive treatment for child
* Parent training while intervention period
* Planed start, change or discontinuation of psychopharmacological treatment for child while intervention period
* No parental adherence or willingness for randomisation process
* Language or reading difficulties of participating parent

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change Oppositional Defiant Disorder subscale score of the Symptom Checklist Disruptive Behavior Disorder (SCL-ODD; Döpfner, Görtz-Dorten, & Lehmkuhl, 2008) | pre, intermediate, post, 6-month FU, 12-month FU
  Questionnaire considers the diagnostic criteria of DSM-IV and ICD-10 for ODD. Informant is participating parent.
Change total score of the Symptom Checklist Attention-Deficit/Hyperactivity Disorder (SCL-ADHD; Döpfner, Görtz-Dorten, & Lehmkuhl, 2008) | pre, intermediate, post, 6-month FU, 12-month FU
  Questionnaire considers the diagnostic criteria of DSM-IV and ICD-10 for ADHD. Informant is participating parent.
Change Oppositional Defiant Disorder subscale score of the Diagnostic Checklist Disruptive Behavior Disorder (DCL-ODD; Döpfner, Görtz-Dorten, & Lehmkuhl, 2008) | pre, intermediate, post, 6-month FU, 12-month FU
  Diagnostic interview considers the criteria of DSM-IV and ICD-10 for ODD. Informant is mental health worker.
Change total score of the Diagnostic Checklist Attention-Deficit/Hyperactivity Disorder (DCL-ADHD; Döpfner, Görtz-Dorten, & Lehmkuhl, 2008) | pre, intermediate, post, 6-month FU, 12-month FU
  Diagnostic interview considers the criteria of DSM-IV and ICD-10 for ADHD. Informant is mental health worker.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Döpfner, PhD, Principal Investigator — University of Cologne
Locations (1):
- Department of Child and Adolescent Psychiatry and Psychotherapy at the University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Hautmann C, Dose C, Hellmich M, Scholz K, Katzmann J, Pinior J, Gebauer S, Nordmann L, Wolff Metternich-Kaizman T, Schurmann S, Dopfner M. Behavioural and nondirective parent training for children with externalising disorders: First steps towards personalised treatment recommendations. Behav Res Ther. 2023 Apr;163:104271. doi: 10.1016/j.brat.2023.104271. Epub 2023 Feb 1. PMID 36931110
- [Derived] Treier AK, Hautmann C, Dose C, Nordmann L, Katzmann J, Pinior J, Scholz KK, Dopfner M. Process Mechanisms in Behavioral Versus Nondirective Guided Self-help for Parents of Children with Externalizing Behavior. Child Psychiatry Hum Dev. 2024 Apr;55(2):453-466. doi: 10.1007/s10578-022-01400-0. Epub 2022 Sep 6. PMID 36064990
- [Derived] Treier AK, Hautmann C, Katzmann J, Nordmann L, Pinior J, Scholz KK, Dopfner M. Treatment components in behavioral versus nondirective telephone-assisted self-help interventions for parents of children with externalizing behavior problems. J Clin Psychol. 2022 May;78(5):735-746. doi: 10.1002/jclp.23255. Epub 2021 Sep 24. PMID 34560813
- [Derived] Del Giudice T, Tervoort J, Hautmann C, Walter D, Dopfner M. Cross-Cultural Validity of the Child and Adolescent Dispositions Model in a Clinical Sample of Children With Externalizing Behavior Problems. Front Psychol. 2020 Apr 8;11:641. doi: 10.3389/fpsyg.2020.00641. eCollection 2020. PMID 32322227